CLINICAL TRIAL: NCT06443879
Title: Loss and Return of Sensation After Axillary Brachial Plexus Nerve Block - Distally or Proximally
Acronym: LRNB
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: W1049
Record Dates: First submitted 2024-03-23; First posted 2024-06-05 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-09

CONDITIONS: Anesthesia
Keywords: Peripheral regional anesthesia; Loss and return of sensation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Axillary brachial plexus nerve block: loss and return of sensation — Evaluating loss and return of sensation after axillary brachial plexus nerve block

SUMMARY:
Peripheral regional anesthesia is the current gold standard of opioid-sparing perioperative analgesia, especially in shoulder, upper limb, and leg surgery. Axillary brachial plexus nerve block is one possible block for upper limb surgery. Loss and return of sensation require time and loss of sensation is supposed to spread from the proximal part to the distal part of the upper limb. Interestingly, until now there is no study about the return of sensation related to the anatomic region.

The investigators hypothesize that the loss and return of sensation after axillary brachial plexus nerve block will first occur in the proximal part of the upper limb and last in the distal part.

DETAILED DESCRIPTION:
Peripheral regional anesthesia is the current gold standard of opioid-sparing perioperative analgesia, especially in shoulder, upper limb, and leg surgery.(1-8) Axillary brachial plexus nerve block is one possible block for upper limb surgery.(4, 5, 9) Loss and return of sensation require time. It is known from clinical practice that loss of sensation occurs from the proximal part of the arm to the distal part of the upper limb.

Interestingly, until now there is no study about the return of sensation related to the anatomic region. The investigators hypothesize that return of sensation after axillary brachial plexus nerve block will develop in the same direction like loss of sensation, what means from proximal to the distal part of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with planed surgery with axillary brachial plexus nerve block
* Informed consent as documented by signature
* Age ≥ 18 years

Exclusion Criteria:

* Patients with a known allergy towards the local anaesthetic

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All outpatients undergoing upper limb surgery with axillary brachial plexus nerve block at Balgrist University Hospital will be eligible to take part in the project.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Loss of sensation after axillary brachial plexus nerve block | Pre-surgery
  A questionnaire will be used to record the loss of sensation in the upper limb. Sensation loss is recorded separately for the finger, hand, forearm, elbow, and arm. It will distinguish between initial and complete loss of sensation.
Return of sensation after axillary brachial plexus nerve block | Immediately after the surgery
  A questionnaire will be used to record the return of sensation in the upper limb. Sensation return is recorded separately for the finger, hand, forearm, elbow, and arm. It will distinguish between initial and complete return of sensation.

SECONDARY OUTCOMES:
Pain before | Pre-surgery
  Pain score (Numeric Rating Scale: 0 to 10) before loss of sensation after the axillary brachial plexus nerve block on a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Pain after | Immediately after the surgery
  Pain score (Numeric Rating Scale: 0 to 10) after loss of sensation after the axillary brachial plexus nerve block on a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable.
Block failure | Pre-surgery
  Block failure yes or no
Amount of pain medication | Immediately after the surgery up to 2 days
  Amount of pain medication after surgery, measured in mg
Prolongation of hospitalization | Immediately after the surgery
  The patient is expected to be an outpatient. If this does not occur, the days of hospitalization will be recorded.
Patients satisfaction with pain therapy | Immediately after the surgery
  The patient will be asked to rate their satisfaction with the pain therapy on a scale from 0 to 10, with 0 indicating very dissatisfied and 10 indicating very satisfied.
Satisfaction of medical staff with the execution of the axillary brachial plexus nerve block | Immediately after the surgery
  The medical staff will be asked to rate their satisfaction with the execution of the axillary brachial plexus nerve block on a scale from 0 to 10, with 0 indicating very dissatisfied and 10 indicating very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Hagen Bomberg, Dr.med., Principal Investigator — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bomberg H, Bayer I, Wagenpfeil S, Kessler P, Wulf H, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Spies C, Kutter B, Winckelmann J, Liebl-Biereige S, Meissner W, Vicent O, Koch T, Sessler DI, Volk T, Raddatz A. Prolonged Catheter Use and Infection in Regional Anesthesia: A Retrospective Registry Analysis. Anesthesiology. 2018 Apr;128(4):764-773. doi: 10.1097/ALN.0000000000002105. PMID 29420315
- [Background] Bomberg H, Huth A, Wagenpfeil S, Kessler P, Wulf H, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Spies C, Kutter B, Winckelmann J, Burgard G, Vicent O, Koch T, Sessler DI, Volk T, Raddatz A. Psoas Versus Femoral Blocks: A Registry Analysis of Risks and Benefits. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):719-724. doi: 10.1097/AAP.0000000000000643. PMID 28806216
- [Background] Bomberg H, Kubulus C, List F, Albert N, Schmitt K, Graber S, Kessler P, Steinfeldt T, Standl T, Gottschalk A, Wirtz SP, Burgard G, Geiger P, Spies CD, Volk T; German Network for Regional Anaesthesia Investigators. Diabetes: a risk factor for catheter-associated infections. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):16-21. doi: 10.1097/AAP.0000000000000196. PMID 25474624
- [Background] Bomberg H, Lorenzana D, Aguirre J, Eichenberger U. [Peripheral Regional Anaesthesia for Perioperative Analgesia]. Praxis (Bern 1994). 2021 Aug;110(10):579-589. doi: 10.1024/1661-8157/a003682. German. PMID 34344186
- [Background] Bomberg H, Wetjen L, Wagenpfeil S, Schope J, Kessler P, Wulf H, Wiesmann T, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Kutter B, Winckelmann J, Liebl-Biereige S, Meissner W, Vicent O, Koch T, Burkle H, Sessler DI, Volk T. Risks and Benefits of Ultrasound, Nerve Stimulation, and Their Combination for Guiding Peripheral Nerve Blocks: A Retrospective Registry Analysis. Anesth Analg. 2018 Oct;127(4):1035-1043. doi: 10.1213/ANE.0000000000003480. PMID 29863605
- [Background] Donauer K, Bomberg H, Wagenpfeil S, Volk T, Meissner W, Wolf A. Regional vs. General Anesthesia for Total Knee and Hip Replacement: An Analysis of Postoperative Pain Perception from the International PAIN OUT Registry. Pain Pract. 2018 Nov;18(8):1036-1047. doi: 10.1111/papr.12708. Epub 2018 Jun 25. PMID 29758587
- [Background] Gabriel RA, Swisher MW, Sztain JF, Furnish TJ, Ilfeld BM, Said ET. State of the art opioid-sparing strategies for post-operative pain in adult surgical patients. Expert Opin Pharmacother. 2019 Jun;20(8):949-961. doi: 10.1080/14656566.2019.1583743. Epub 2019 Feb 27. PMID 30810425
- [Background] Luedi MM, Upadek V, Vogt AP, Steinfeldt T, Eichenberger U, Sauter AR. A Swiss nationwide survey shows that dual guidance is the preferred approach for peripheral nerve blocks. Sci Rep. 2019 Jun 24;9(1):9178. doi: 10.1038/s41598-019-45700-3. PMID 31235760
- [Background] Marhofer P, Eichenberger U, Stockli S, Huber G, Kapral S, Curatolo M, Kettner S. Ultrasonographic guided axillary plexus blocks with low volumes of local anaesthetics: a crossover volunteer study. Anaesthesia. 2010 Mar;65(3):266-71. doi: 10.1111/j.1365-2044.2010.06247.x. Epub 2010 Jan 29. PMID 20121770